CLINICAL TRIAL: NCT05234567
Title: A Prospective Observational Sub-Study of the Global Hypophosphatasia Registry to Describe the Potential Risk of Immune-Mediated Loss of Pharmacological Effect of Asfotase Alfa in Participants With Hypophosphatasia
Brief Title: A Prospective Sub-Study of the Global Hypophosphatasia Registry
Status: Recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-HPP-501s
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hypophosphatasia
Keywords: Pediatric Onset; HPP; Asfotase alfa
MeSH Terms: conditions — Hypophosphatasia | interventions — asfotase alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Pediatric-onset HPP: Each participant will be followed for a minimum of 5 years or, if applicable, until early withdrawal. Biochemical, clinical, imaging (if clinically indicated), and functional/quality of life outcomes relevant to HPP will be assessed.
  Interventions: Biological: Asfotase Alfa

INTERVENTIONS:
Biological: Asfotase Alfa — All participants will receive asfotase alfa subcutaneously per standard of care. Unless otherwise specified per the Physician's standard of care, participants aged < 2 years are recommended for a clinic visit approximately every 3 months after Enrollment until 2 years of age, after which they should have a clinic visit approximately every 6 months. Participants should be followed for 5 years, as possible.
  Other Names: Strensiq

SUMMARY:
In this prospective observational sub-study, participants with pediatric-onset hypophosphatasia (HPP) (perinatal/infantile- or juvenile-onset) of any age will be followed for a minimum of 5 years at sites in the United States and potentially 1 or 2 other countries.

ELIGIBILITY:
Inclusion Criteria:

* Any age or sex with a confirmed diagnosis of pediatric-onset HPP (that is, first HPP sign or symptom presented at < 18 years of age).
* Currently receiving asfotase alfa treatment at Enrollment (not treatment-naïve) or the Physician has decided to resume (not treatment-naïve) or start (treatment-naïve) the participant's asfotase alfa treatment within 6 months after Enrollment.
* Participant must have documented alkaline phosphatase (ALP) activity below the lower limit of normal for age and sex, and a documented ALPL gene mutation (Note: An exception is made for infants with clinical features of HPP plus low ALP who need to start asfotase alfa treatment right away, at the Physician's discretion, but do not yet have a genetic result. In this case, ALPL gene documentation is not required at the time of sub-study enrollment but should be documented within 6 months after Enrollment).
* Participant or participant's parent/legally authorized representative is able to read and/or understand the informed consent and study questionnaires in the local language.
* Participant or participant's parent/legally authorized representative must be willing and able to give signed informed consent for this sub-study, and the participant must be willing to give written informed assent, if appropriate and required by local regulations.

Exclusion Criteria:

* Currently participating in an Alexion-sponsored interventional clinical study. Participants who have concluded participation in an Alexion-sponsored asfotase alfa clinical study are eligible to enroll in this sub-study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HPP
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2028-07-18 (Estimated); Study Completion 2028-07-18 (Estimated)

PRIMARY OUTCOMES:
Occurrence Of Immune-mediated Loss Of Effectiveness According To The Treating Physician | Up to 5 years
  This will be based on clinical and biochemical assessments as well as positive anti-drug antibodies and positive neutralizing antibodies.
Occurrence Of Immune-mediated Serious Adverse Events | Up to 5 years
  These serious adverse events will include serious hypersensitivity reactions and anaphylaxis.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Clinical Trial Site, Hartford, Connecticut
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Kansas City, Missouri
  - Clinical Trial Site, Mineola, New York
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Salt Lake City, Utah
  - Clinical Trial Site, Charlottesville, Virginia
  - Clinical Trial Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: Alexion will consider requests for disclosure of clinical study participant-level data provided that participant privacy is assured through methods like data de-identification, pseudonymization, or anonymization (as required by applicable law), and if such disclosure was included in the relevant study informed consent form or similar documentation. Qualified academic investigators may request participant-level clinical data and supporting documents (statistical analysis plan and protocol) pertaining to Alexion-sponsored studies. Further details regarding data availability and instructions for requesting information are available in the Alexion Clinical Trials Disclosure and Transparency Policy at https://alexion.com/our-research/research-and-development.